CLINICAL TRIAL: NCT03284957
Title: A Phase 1/2 Study for the Safety, Efficacy, Pharmacokinetic and Pharmacodynamics Evaluation of Amcenestrant (SAR439859), Administered Orally as Monotherapy, Then in Combination With Other Anti-cancer Therapies in Postmenopausal Women With Estrogen Receptor-positive Advanced Breast Cancer
Brief Title: Phase 1/2 Study of Amcenestrant (SAR439859) Single Agent and in Combination With Other Anti-cancer Therapies in Postmenopausal Women With Estrogen Receptor Positive Advanced Breast Cancer
Acronym: AMEERA-1
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision to prematurely stop the study, not linked to any safety concern.
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TED14856; U1111-1189-4896 (Registry Identifier: ICTRP); 2024-512997-89 (Registry Identifier: CTIS); 2017-000690-36 (EudraCT Number)
Record Dates: First submitted 2017-09-13; First posted 2017-09-15 (Actual); Results first posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib; Alpelisib; Everolimus; abemaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Amcenestrant Monotherapy: Arm #1 Part A Dose Escalation, Part B Dose Expansion (Experimental): Part A: Amcenestrant will be administered orally once daily (QD). Treatment will begin with an identified starting dose. Administration of higher doses to subsequent participants is based on occurrence of DLTs and evaluation of target saturation and PK parameters at initial and subsequent doses, until maximum administered dose (MAD) is reached. Drug will be administered in a 28-day cycle.
  Part B: When the dose escalation phase ends, the recommended dose will be administered for the expansion cohort. Drug will be administered in a 28-day cycle.
  Interventions: Drug: Amcenestrant
- Amcenestrant/Palbociclib: Arm #2 Part C Dose Escalation, Part D Dose Expansion (Experimental): Part C: Amcenestrant will be administered in combination with palbociclib: amcenestrant starting oral daily dose will be one dose level below monotherapy RD and palbociclib will be dosed at fixed standard dose. Administration of higher dose of amcenestrant (with standard palbociclib dose) to subsequent participants will be based on occurrence of DLTs at initial and subsequent doses, until MAD of amcenestrant is reached. Drugs will be administered in a 28-day cycle (palbociclib will be administered for 21 days of cycle).
  Part D: Based on the results in Part C, participants will be administered either: 1) a determined amcenestrant dose (RD) with standard dose of palbociclib in combination therapy, or 2) one of two randomized dose levels of amcenestrant with standard dose of palbociclib in combination therapy. Drugs will be administered in a 28-day cycle (palbociclib will be administered for 21 days of cycle).
  Interventions: Drug: Amcenestrant; Drug: Palbociclib
- Amcenestrant/Alpelisib: Arm #3 Part F Safety Run-In, Part G Dose Expansion (Experimental): Part F: Amcenestrant will be administered in combination with alpelisib at a fixed standard dose. Additional dose levels of amcenestrant with alpelisib could be explored if needed based on the safety and PK results. Lower dose of alpelisib could be explored based on the PK results and safety profile from the initial combination administration. Both amcenestrant and alpelisib will be administered in a 28-day cycle.
  Part G: Based on the conclusion in Part F, participants will be administered the determined RD of amcenestrant and alpelisib given in the combination in an expansion cohort. Both study drugs will be administered in a 28-day cycle.
  Interventions: Drug: Amcenestrant; Drug: Alpelisib
- Amcenestrant/Everolimus: Arm #4 Part H Dose Escalation, Part I Dose Expansion (Experimental): Part H: Amcenestrant will be administered at the determined RD in combination with 2 dose levels of everolimus. Additional dose levels of amcenestrant with everolimus could be explored if needed based on the safety and PK results. Both amcenestrant and everolimus will be administered in a 28-day cycle.
  Part I: Based on the conclusion in Part H, participants will be administered the determined RD of amcenestrant and RD of everolimus given in the combination in an expansion cohort. Both study drugs will be administered in a 28-day cycle.
  Interventions: Drug: Amcenestrant; Drug: Everolimus
- Amcenestrant/Abemaciclib: Arm #5 Part J Dose Escalation, Part K Dose Expansion (Experimental): Part J: Amcenestrant will be administered at the determined RD in combination with 2 dose levels of abemaciclib. Additional dose levels of amcenestrant with abemaciclib could be explored if needed based on the safety and PK results. Both amcenestrant and abemaciclib will be administered in a 28-day cycle.
  Part K: Based on the conclusion in Part J, participants will be administered the determined RD of amcenestrant and RD of abemaciclib given in the combination in an expansion cohort. Both study drugs will be administered in a 28-day cycle.
  Interventions: Drug: Amcenestrant; Drug: Abemaciclib

INTERVENTIONS:
Drug: Amcenestrant — Pharmaceutical form: capsule
  Route of administration: oral
  Other Names: SAR439859
Drug: Palbociclib — Pharmaceutical form: capsule
  Route of administration: oral
  Other Names: Ibrance®
  Arms: Amcenestrant/Palbociclib: Arm #2 Part C Dose Escalation, Part D Dose Expansion
Drug: Alpelisib — Pharmaceutical form: tablet
  Route of administration: oral
  Other Names: Piqray®
  Arms: Amcenestrant/Alpelisib: Arm #3 Part F Safety Run-In, Part G Dose Expansion
Drug: Everolimus — Pharmaceutical form: tablet
  Arms: Amcenestrant/Everolimus: Arm #4 Part H Dose Escalation, Part I Dose Expansion
Drug: Abemaciclib — Pharmaceutical form: tablet
  Other Names: Verzenio®
  Arms: Amcenestrant/Abemaciclib: Arm #5 Part J Dose Escalation, Part K Dose Expansion

SUMMARY:
Primary Objectives:

Dose Escalation:

* To assess the incidence rate of dose-limiting toxicity (DLT) and to determine the maximum tolerated dose (MTD) as well as the recommended dose (RD) of amcenestrant administered as monotherapy and in combination with palbociclib
* To assess the incidence rate of DLT and determine the RD of everolimus or abemaciclib in combination with the selected amcenestrant dose for the combination therapy

Safety Run-In:

- To confirm the RD of amcenestrant in combination with alpelisib

Dose Expansion:

* Antitumor activity using objective response rate (ORR)
* Overall safety profile of amcenestrant administered in combination with palbociclib, alpelisib, everolimus, and abemaciclib

Secondary Objectives:

* Overall safety profile of amcenestrant monotherapy and in combination
* Pharmacokinetic (PK) profile of amcenestrant administered as monotherapy or in combination and PK profile of palbociclib, alpelisib, everolimus and abemaciclib
* Antitumor activity using ORR, the clinical benefit rate (CBR) and progression free survival (PFS)
* Time to first tumor response
* Residual ER availability with positron emission tomography (PET) scan [(18)F] fluoroestradiol (18F-FES) uptake with increasing doses of amcenestrant
* Food effect on PK of amcenestrant
* Potential induction/inhibition effect of amcenestrant on cytochrome P450 (CYP) 3A using 4b-OH cholesterol

DETAILED DESCRIPTION:
Duration of the study, per participant, will include eligibility period (screening period) of up to 4 weeks (28 days), treatment period (at least 1 cycle [28 days] of study treatment), and end of treatment (EOT) visit at least 22 to 30 days (or until the participant receives another anticancer therapy, whichever is earlier) following the last study treatment administration. The expected enrollment period is approximately 60 months.

ELIGIBILITY:
Inclusion criteria:

* Participants must be postmenopausal women
* Histological diagnosis of breast adenocarcinoma
* Locally advanced or metastatic disease
* Either primary tumor or any metastatic site to be positive for Estrogen Receptors (ER+) and negative for HER2 (HER2-) receptor
* Participants must have been previously treated with at least 6 months of endocrine therapy for advanced disease:
* Dose Escalation study parts:

Arm #3 - Part F and Arm #5 - Part J: up to 2 prior lines of either single endocrine therapy and/or endocrine-based therapy Arm #4 -H: up to 2 prior lines of either single endocrine therapy and/or endocrine-based therapy (exemestane not allowed)

- Dose Expansion study parts: Arm #2: - Part D: no more than 2 prior lines of advanced endocrine therapy for advanced disease are allowed Arm #3, - Part G: patients must have received and progressed on the combination of Aromatase Inhibitors (AI) + CDK4/6 inhibitor as the first line (1L) treatment for advanced disease Arm #4 - Part I: participants must have received and progressed on the combination of Aromatase Inhibitors (AI) +CDK4/6 Inhibitor as the first line (1L) treatment for advanced disease (exemestane not allowed) Arm#5: - Part K: up to 1 prior line of a single endocrine therapy for advanced disease Note: Additional patients who relapsed while on previous adjuvant endocrine therapy that was initiated ≥24 months ago, or relapsed < 12 months after completion of adjuvant endocrine therapy are also allowed for Arms #2, #3, #4, and #5 (Parts C, D, F, G, H, I, J and K).

* Participants previously treated with chemotherapy for advanced disease: no more than 3 prior chemotherapeutic regimens in Arm #1 Part A, and no more than 1 prior chemotherapeutic regimen in Arms #1, #2, #3, #4, and #5 (Parts B, C, D, F, H and J respectively); prior chemotherapy for advanced disease is not allowed in dose expansion of Arms #3, #4, and #5 (Part G, I and K respectively).
* Measurable lesion

Exclusion criteria:

* Medical history or ongoing gastrointestinal disorders that could affect absorption of oral study drugs (including difficulties with swallowing capsules)
* Participants with any other cancer (except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer or any other cancer from which the participant has been disease free for >3 years)
* Participants with known brain metastases
* Treatment with anticancer agents (including investigational drugs) less than 2 weeks before first study treatment starts (less than 4 weeks if the anticancer agents were antibodies)
* Prior treatment with another selective ER down-regulator (SERD)
* Dose Escalation study parts (Parts F, H and J): SERDs are not allowed except for fulvestrant which will need a washout of at least 6 weeks prior to the first study drug administration
* Dose Expansion study parts (Parts G, I and K): prior (last) treatment with any SERD including fulvestrant will not be allowed
* Inadequate hematological and biochemical lab tests
* Participants with Gilbert disease
* Treatment with HIV-antiviral, antifungal and antioxidant agents less than 2 weeks before study treatment starts
* Treatment with strong P450 (CYP) 3A inducers within 2 weeks before first study treatment
* Treatment with OATP1B1/B3 sensitive substrates and which cannot be replaced
* Arm#2 Treatment with strong CYP3A inhibitors within 2 weeks before first study treatment starts
* More than one prior advanced cyclin-dependent kinase (CDK) 4/6 inhibitor-based therapy in Arm #1, Arm #2 (Part C), Arm #3 (Parts F and G), and Arm#4 (Part H).
* Arm #2, #3, #4 and #5 (Parts C, D, F, G, H, I, J and K) only: participants with concurrent or history of pneumonitis
* Arm #3, #4 and #5 (Parts F, G, H, I, J and K) only: prior treatment therapies that target the PI3K axis (mTOR inhibitors, AKT inhibitors, PI3K inhibitors)
* Arm #3 and #4 (Parts F, G, H and I) only: participants with diabetes mellitus type-I or uncontrolled diabetes mellitus type-II: ie, fasting plasma glucose ≥ 140mg/dl (7.7 mmol/l) or HbA1C > 6.2%
* Arm #3 and #4 (Parts F, G, H and I) only: history of severe cutaneous reaction (eg. Stevens-Johnson syndrome [SJS], erythema multiforme [EM]), toxic epidermal necrolysis (TEN), and drug reaction with eosinophilia and systemic symptoms [DRESS].
* Arm #3 (Parts F and G) only: ongoing osteonecrosis of jaw
* Arm #4 (Parts H and I) only: any active, untreated or uncontrolled infection (e.g. viral, bacterial, fungal etc.)
* Arm #4 (Parts H and I) only: participants with active and uncontrolled stomatitis, angioedema due to concomitant treatment with ACE inhibitors, impaired wounds
* Arm #4 (Parts H and I) only: uncontrolled hypercholesterolemia, hypertriglyceridemia and hyperglycemia in non-diabetic participants
* Arm #4 (Parts H and I) only: treatment with strong or moderate CYP3A4 inhibitors, strong CYP3A4 inducers and/or P-gp inhibitors within 2 weeks before the first study treatment administration or 5 elimination half-lives, whichever is the longest
* Arm #5 (Parts J and K) only: history or current (controlled/not controlled) venous thromboembolism (i.e. deep vein thrombosis (DVT), pulmonary embolism (PE), cerebral venous sinus thrombosis (CVST)

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2024-11-08 (Actual); Study Completion 2024-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (25):
- United States (4):
  - University of Colorado - Anschutz Medical Campus- Site Number : 8400005, Aurora, Colorado
  - Massachusetts General Hospital- Site Number : 8400002, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center - New York - York Avenue- Site Number : 8400003, New York, New York
  - Fred Hutchinson Cancer Center- Site Number : 8400001, Seattle, Washington
- Investigational Site Number : 0560001, Leuven, Belgium
- Canada (3):
  - Investigational Site Number : 1240004, Edmonton, Alberta
  - Investigational Site Number : 1240003, Vancouver, British Columbia
  - Investigational Site Number : 1240002, Toronto, Ontario
- Czechia (3):
  - Investigational Site Number : 2030002, Brno
  - Investigational Site Number : 2030001, Prague
  - Investigational Site Number : 2030003, Prague
- France (5):
  - Investigational Site Number : 2500002, Bordeaux
  - Investigational Site Number : 2500005, Lille
  - Investigational Site Number : 2500003, Lyon
  - Investigational Site Number : 2500001, Saint-Herblain
  - Investigational Site Number : 2500004, Villejuif
- Investigational Site Number : 3800003, Milan, Milano, Italy
- Investigational Site Number : 6160004, Gdynia, Pomeranian Voivodeship, Poland
- Portugal (2):
  - Investigational Site Number : 6200001, Lisbon
  - Investigational Site Number : 6200002, Lisbon
- Spain (3):
  - Investigational Site Number : 7240007, Madrid
  - Investigational Site Number : 7240001, Madrid
  - Investigational Site Number : 7240002, Madrid
- United Kingdom (2):
  - Investigational Site Number : 8260002, Cardiff, Cardiff [Caerdydd Gb-crd]
  - Investigational Site Number : 8260003, Oxford, Oxfordshire

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Bardia A, Chandarlapaty S, Linden HM, Ulaner GA, Gosselin A, Cartot-Cotton S, Cohen P, Doroumian S, Paux G, Celanovic M, Pelekanou V, Ming JE, Ternes N, Bouaboula M, Lee JS, Bauchet AL, Campone M. AMEERA-1 phase 1/2 study of amcenestrant, SAR439859, in postmenopausal women with ER-positive/HER2-negative advanced breast cancer. Nat Commun. 2022 Jul 15;13(1):4116. doi: 10.1038/s41467-022-31668-8. PMID 35840573
- See also: TED14856 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=26150&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 25 sites in 10 countries between 20-Sep-2017 and 08-Nov-2024. A total of 136 participants were enrolled in the study. Sponsor decided to prematurely stop the study, it was not linked to any safety concern.
Pre-assignment Details: The study consisted of dose-escalation phases (Parts A, C, H, J), safety run-in phase (Part F) and dose-expansion phases (Parts B, D, G, I, K). Participants received amcenestrant as monotherapy (Parts A, B) or in combination with palbociclib (Parts C, D), alpelisib (Part F), everolimus (Parts H, I) or abemaciclib (Part J). Parts G and K were never initiated due to the early termination of the study. Reason for not completed = reason for permanent full treatment discontinuation.
Groups:
- Part A: Amcenestrant 20 mg: Participants received amcenestrant 20 milligrams (mg) capsule orally once daily (QD) in a fasted state (no dose on Cycle 1 Day 2, dose administered in a fed state on Cycle 1 Day 3 only) in 28-day cycles until disease progression, unacceptable toxicity, participant's wish to stop the study, or any other reason, whichever came first.
- Part A: Amcenestrant 150 mg: Participants received amcenestrant 150 mg capsule orally QD in a fasted state (no dose on Cycle 1 Day 2, dose administered in a fed state on Cycle 1 Day 3 only) in 28-day cycles until disease progression, unacceptable toxicity, participant's wish to stop the study, or any other reason, whichever came first.
- Part A: Amcenestrant 200 mg: Participants received amcenestrant 200 mg capsule orally QD in a fasted state (no dose on Cycle 1 Day 2, dose administered in a fed state on Cycle 1 Day 3 only) in 28-day cycles until disease progression, unacceptable toxicity, participant's wish to stop the study, or any other reason, whichever came first.
- Part A: Amcenestrant 400 mg: Participants received amcenestrant 400 mg capsule orally QD in a fasted state (no dose on Cycle 1 Day 2, dose administered in a fed state on Cycle 1 Day 3 only) in 28-day cycles until disease progression, unacceptable toxicity, participant's wish to stop the study, or any other reason, whichever came first.
- Part A: Amcenestrant 600 mg: Participants received amcenestrant 600 mg capsule orally QD in a fasted state (no dose on Cycle 1 Day 2, dose administered in a fed state on Cycle 1 Day 3 only) in 28-day cycles until disease progression, unacceptable toxicity, participant's wish to stop the study, or any other reason, whichever came first.
- Part A: Amcenestrant 300 mg BID: Participants received amcenestrant 300 mg capsule orally once on Cycle 1 Day 1 and then twice daily (BID) from Cycle 1 Day 3 onwards (no dose on Cycle 1 Day 2) in a fed or fasted state in 28-day cycles until disease progression, unacceptable toxicity, participant's wish to stop the study, or any other reason, whichever came first.
- Part B: Amcenestrant 400 mg: Participants received amcenestrant 400 mg capsule orally QD in a fed or fasted state in 28-day cycles until disease progression, unacceptable toxicity, participant's wish to stop the study, or any other reason, whichever came first.
- Part C: Amcenestrant 200 mg + Palbociclib 125 mg; Part D: Amcenestrant 200 mg + Palbociclib 125 mg: Participants received amcenestrant 200 mg capsule orally QD in a fed state along with palbociclib 125 mg capsule orally QD in a fed state for 21 consecutive days followed by 7 days off treatment in 28-day cycles until disease progression, unacceptable toxicity, participant's wish to stop the study, or any other reason, whichever came first.
- Part C: Amcenestrant 400 mg + Palbociclib 125 mg: Participants received amcenestrant 400 mg capsule orally QD in a fed state along with palbociclib 125 mg capsule orally QD in a fed state for 21 consecutive days followed by 7 days off treatment in 28-day cycles until disease progression, unacceptable toxicity, participant's wish to stop the study, or any other reason, whichever came first.
- Part F: Amcenestrant 200 mg + Alpelisib 300 mg: Participants received amcenestrant 200 mg capsule orally QD in a fed state from Cycle 1 Day 4 onwards along with alpelisib 300 mg tablet orally QD in a fed state in 28-day cycles until disease progression, unacceptable toxicity, participant's wish to stop the study, or any other reason, whichever came first.
- Part H: Amcenestrant 200 mg + Everolimus 5 mg: Participants received amcenestrant 200 mg capsule orally QD in a fed state along with everolimus 5 mg tablet orally QD in a fed state in 28-day cycles until disease progression, unacceptable toxicity, participant's wish to stop the study, or any other reason, whichever came first.
- Part H: Amcenestrant 200 mg + Everolimus 10 mg; Part I: Amcenestrant 200 mg + Everolimus 10 mg: Participants received amcenestrant 200 mg capsule orally QD in a fed state along with everolimus 10 mg tablet orally QD in a fed state in 28-day cycles until disease progression, unacceptable toxicity, participant's wish to stop the study, or any other reason, whichever came first.
- Part J: Amcenestrant 200 mg + Abemaciclib 100 mg BID: Participants received amcenestrant 200 mg capsule orally QD in a fed state along with abemaciclib 100 mg tablet orally BID in a fed state in 28-day cycles until disease progression, unacceptable toxicity, participant's wish to stop the study, or any other reason, whichever came first.
- Part J: Amcenestrant 200 mg + Abemaciclib 150 mg BID: Participants received amcenestrant 200 mg capsule orally QD in a fed state along with abemaciclib 150 mg tablet orally BID in a fed state in 28-day cycles until disease progression, unacceptable toxicity, participant's wish to stop the study, or any other reason, whichever came first.
Period: Overall Study
Arm/Group | Part A: Amcenestrant 20 mg | Part A: Amcenestrant 150 mg | Part A: Amcenestrant 200 mg | Part A: Amcenestrant 400 mg | Part A: Amcenestrant 600 mg | Part A: Amcenestrant 300 mg BID | Part B: Amcenestrant 400 mg | Part C: Amcenestrant 200 mg + Palbociclib 125 mg | Part C: Amcenestrant 400 mg + Palbociclib 125 mg | Part D: Amcenestrant 200 mg + Palbociclib 125 mg | Part F: Amcenestrant 200 mg + Alpelisib 300 mg | Part H: Amcenestrant 200 mg + Everolimus 5 mg | Part H: Amcenestrant 200 mg + Everolimus 10 mg | Part I: Amcenestrant 200 mg + Everolimus 10 mg | Part J: Amcenestrant 200 mg + Abemaciclib 100 mg BID | Part J: Amcenestrant 200 mg + Abemaciclib 150 mg BID
Started | 3 | 3 | 4 | 3 | 3 | 6 | 49 | 9 | 6 | 30 | 8 | 3 | 3 | 1 | 3 | 2
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 4 | 3 | 3 | 6 | 49 | 9 | 6 | 30 | 8 | 3 | 3 | 1 | 3 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 4 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 3 | 3 | 4 | 3 | 3 | 5 | 45 | 8 | 5 | 18 | 7 | 2 | 3 | 1 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 6 | 0 | 0 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: The safety population included all registered participants exposed to the study treatment, regardless of the amount of treatment administered.
Groups:
- Part A: Amcenestrant 20 mg: Participants received amcenestrant 20 mg capsule orally QD in a fasted state (no dose on Cycle 1 Day 2, dose administered in a fed state on Cycle 1 Day 3 only) in 28-day cycles until disease progression, unacceptable toxicity, participant's wish to stop the study, or any other reason, whichever came first.
- Part A: Amcenestrant 300 mg BID: Participants received amcenestrant 300 mg capsule orally once on Cycle 1 Day 1 and then BID from Cycle 1 Day 3 onwards (no dose on Cycle 1 Day 2) in a fed or fasted state in 28-day cycles until disease progression, unacceptable toxicity, participant's wish to stop the study, or any other reason, whichever came first.
- Total: Total of all reporting groups
Arm/Group | Part A: Amcenestrant 20 mg | Part A: Amcenestrant 150 mg | Part A: Amcenestrant 200 mg | Part A: Amcenestrant 400 mg | Part A: Amcenestrant 600 mg | Part A: Amcenestrant 300 mg BID | Part B: Amcenestrant 400 mg | Part C: Amcenestrant 200 mg + Palbociclib 125 mg | Part C: Amcenestrant 400 mg + Palbociclib 125 mg | Part D: Amcenestrant 200 mg + Palbociclib 125 mg | Part F: Amcenestrant 200 mg + Alpelisib 300 mg | Part H: Amcenestrant 200 mg + Everolimus 5 mg | Part H: Amcenestrant 200 mg + Everolimus 10 mg | Part I: Amcenestrant 200 mg + Everolimus 10 mg | Part J: Amcenestrant 200 mg + Abemaciclib 100 mg BID | Part J: Amcenestrant 200 mg + Abemaciclib 150 mg BID | Total
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 6 | 49 | 9 | 6 | 30 | 8 | 3 | 3 | 1 | 3 | 2 | 136
Age, Customized [Count of Participants; unit: Participants]
  From 18 - 64 years | 1 | 3 | 3 | 1 | 3 | 5 | 29 | 6 | 2 | 19 | 4 | 2 | 2 | 1 | 2 | 0 | 83
  From 65 - 84 years | 2 | 0 | 1 | 2 | 0 | 0 | 17 | 3 | 4 | 9 | 4 | 1 | 1 | 0 | 1 | 2 | 47
  85 years and over | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 4 | 3 | 3 | 6 | 49 | 9 | 6 | 30 | 8 | 3 | 3 | 1 | 3 | 2 | 136
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 1 | 3 | 1 | 3 | 2 | 3 | 35 | 4 | 4 | 29 | 6 | 0 | 3 | 0 | 2 | 2 | 98
  Black or African American | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Not reported | 2 | 0 | 2 | 0 | 1 | 2 | 13 | 3 | 2 | 0 | 2 | 3 | 0 | 1 | 1 | 0 | 32
  Unknown | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Parts A, C, F, H, J: Number of Participants With Study Treatment-Related Dose-Limiting Toxicities (DLTs)
Description: DLTs: any treatment-emergent adverse event(TEAE) related to study treatment per National Cancer Institute Common Terminology Criteria for AE scale version (v) 4.03:Grade(G)≥3 nonhematological toxicity except:G3 nausea/vomiting resolved to G≤1 in 48 hours(h),G3 diarrhea with therapy and lasting<48h,G3 hyperglycemia resolved to G≤1 in 48h(Part H);G≥3 hematological toxicity except:G3 anemia,G4 neutropenia<7days(d),G3 neutropenia without fever/infection,G3 thrombocytopenia without bleeding;elevated total serum bilirubin(BL)>2xupper limit of normal(except Part F),Part F:G3 hyperglycemia not resolved to G≤2 in 7d after antidiabetic treatment,G2 hyperglycemia not resolved to G≤1 in 21d,G2 alanine aminotransferase(ALT) increase in conjunction with total blood BL G≥2 without liver metastases,G≥3 ALT/aspartate aminotransferase increase for>4d,G3 rash/maculopapular rash not resolved to G≤1 in 7d;treatment related toxicity causing≥7d omission in Cycle 1 or >2 weeks delay in Cycle 2 in Part C.
Time Frame: Cycle 1 Day 1 to Cycle 1 Day 28 (cycle duration=28 days)
Population: The DLT-evaluable population included participants who received 1 cycle (28 days, oral administration), with intake of at least 75% of intended doses, unless they discontinued study treatment before Cycle 1 completion due to a DLT, and in Part A had an evaluable 18F-fluorestradiol (18F-FES) positron emission tomography (PET) scan at baseline and between Days 11 and 15 of first cycle. Any participant who developed a DLT in Part A despite absence of evaluable 18F-FES-PET scan was also included.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Amcenestrant 20 mg | Part A: Amcenestrant 150 mg | Part A: Amcenestrant 200 mg | Part A: Amcenestrant 400 mg | Part A: Amcenestrant 600 mg | Part A: Amcenestrant 300 mg BID | Part C: Amcenestrant 200 mg + Palbociclib 125 mg | Part C: Amcenestrant 400 mg + Palbociclib 125 mg | Part F: Amcenestrant 200 mg + Alpelisib 300 mg | Part H: Amcenestrant 200 mg + Everolimus 5 mg | Part H: Amcenestrant 200 mg + Everolimus 10 mg | Part J: Amcenestrant 200 mg + Abemaciclib 100 mg BID | Part J: Amcenestrant 200 mg + Abemaciclib 150 mg BID
Number analyzed (Participants) | 3 | 3 | 3 | 2 | 3 | 2 | 9 | 6 | 6 | 3 | 3 | 3 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Part B: Objective Response Rate (ORR) as Determined by Independent Central Review (ICR)
Description: ORR was determined by dividing the number of participants who achieved confirmed complete response (CR) or partial response (PR) by the number of participants from the analysis population. ORR was assessed by ICR according to response evaluation criteria in solid tumors (RECIST) v1.1. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) had a reduction in short axis to <10 millimeters (mm). PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From first dose of study treatment administration (Day 1) up to maximum exposure of study treatment; approximately 278 weeks
Population: The efficacy population included all treated participants with measurable disease at study entry who provided a baseline and at least 1 post-baseline evaluable tumor assessment. Participants with an early progression as per RECIST v1.1 or who died from disease progression were also included in this set.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Part B: Amcenestrant 400 mg
Number analyzed (Participants) | 46
percentage of participants | 10.9 [4.4 to 21.5]

3. Primary Outcome: Parts D, I: Number of Participants With Treatment-Emergent Adverse Events and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: AE was any untoward medical occurrence in a participant or clinical investigation participant administered with a pharmaceutical product and which did not necessarily had a causal relationship with the treatment. SAE was any untoward medical occurrence that at any dose, resulted in death, was life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or was a medically important event. TEAEs were AEs that developed or worsened or became serious during the treatment period.
Time Frame: From first dose of study treatment administration (Day 1) up to 30 days after the last dose of study treatment administration; approximately 232 weeks for Part D and 11 weeks for Part I
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part D: Amcenestrant 200 mg + Palbociclib 125 mg | Part I: Amcenestrant 200 mg + Everolimus 10 mg
Number analyzed (Participants) | 30 | 1
Participants
  TEAEs | 30 | 1
  TESAEs | 8 | 1

4. Secondary Outcome: Parts A, B, C, F, H, J: Number of Participants With Treatment-Emergent Adverse Events and Treatment-Emergent Serious Adverse Events
Description: as for outcome 3
Time Frame: From first dose of study treatment administration (Day 1) up to 30 days after the last dose of study treatment administration; approximately 94, 282, 144, 96, 59, 130 weeks for Parts A, B, C, F, H, J respectively
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Amcenestrant 20 mg | Part A: Amcenestrant 150 mg | Part A: Amcenestrant 200 mg | Part A: Amcenestrant 400 mg | Part A: Amcenestrant 600 mg | Part A: Amcenestrant 300 mg BID | Part B: Amcenestrant 400 mg | Part C: Amcenestrant 200 mg + Palbociclib 125 mg | Part C: Amcenestrant 400 mg + Palbociclib 125 mg | Part F: Amcenestrant 200 mg + Alpelisib 300 mg | Part H: Amcenestrant 200 mg + Everolimus 5 mg | Part H: Amcenestrant 200 mg + Everolimus 10 mg | Part J: Amcenestrant 200 mg + Abemaciclib 100 mg BID | Part J: Amcenestrant 200 mg + Abemaciclib 150 mg BID
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 6 | 49 | 9 | 6 | 8 | 3 | 3 | 3 | 2
Participants
  TEAEs | 3 | 3 | 4 | 3 | 3 | 6 | 49 | 9 | 6 | 8 | 3 | 3 | 3 | 2
  TESAEs | 0 | 1 | 1 | 0 | 1 | 3 | 15 | 2 | 1 | 6 | 1 | 0 | 0 | 1

5. Secondary Outcome: Parts A, B, C, D, F, H, I, J: Objective Response Rate as Determined by Investigators/Local Radiologists
Description: ORR was determined by dividing the number of participants who achieved confirmed CR or PR by the number of participants from the analysis population. ORR was assessed by investigators/local radiologists according to RECIST v1.1. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) had a reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From first dose of study treatment administration (Day 1) up to maximum exposure of study treatment; approximately 90, 278, 140, 228, 92, 55, 7, 126 weeks for Parts A, B, C, D, F, H, I, J respectively
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Part A: Amcenestrant 20 mg | Part A: Amcenestrant 150 mg | Part A: Amcenestrant 200 mg | Part A: Amcenestrant 400 mg | Part A: Amcenestrant 600 mg | Part A: Amcenestrant 300 mg BID | Part B: Amcenestrant 400 mg | Part C: Amcenestrant 200 mg + Palbociclib 125 mg | Part C: Amcenestrant 400 mg + Palbociclib 125 mg | Part D: Amcenestrant 200 mg + Palbociclib 125 mg | Part F: Amcenestrant 200 mg + Alpelisib 300 mg | Part H: Amcenestrant 200 mg + Everolimus 5 mg | Part H: Amcenestrant 200 mg + Everolimus 10 mg | Part I: Amcenestrant 200 mg + Everolimus 10 mg | Part J: Amcenestrant 200 mg + Abemaciclib 100 mg BID | Part J: Amcenestrant 200 mg + Abemaciclib 150 mg BID
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 4 | 46 | 9 | 6 | 29 | 7 | 2 | 3 | 1 | 3 | 2
percentage of participants | 0 [NA to NA] — NA indicates that upper and lower limit of 90% confidence interval (CI) were not estimable due to insufficient number of participants with events. | 33.3 [1.7 to 86.5] | 0 [NA to NA] — NA indicates that upper and lower limit of 90% CI were not estimable due to insufficient number of participants with events. | 0 [NA to NA] — NA indicates that upper and lower limit of 90% CI were not estimable due to insufficient number of participants with events. | 0 [NA to NA] — NA indicates that upper and lower limit of 90% CI were not estimable due to insufficient number of participants with events. | 0 [NA to NA] — NA indicates that upper and lower limit of 90% CI were not estimable due to insufficient number of participants with events. | 8.7 [3.0 to 18.8] | 22.2 [4.1 to 55.0] | 0 [0.0 to 39.3] | 34.5 [20.0 to 51.4] | 0 [NA to NA] — NA indicates that upper and lower limit of 90% CI were not estimable due to insufficient number of participants with events. | 0 [NA to NA] — NA indicates that upper and lower limit of 90% CI were not estimable due to insufficient number of participants with events. | 0 [NA to NA] — NA indicates that upper and lower limit of 90% CI were not estimable due to insufficient number of participants with events. | 0 [NA to NA] — NA indicates that upper and lower limit of 90% CI were not estimable due to insufficient number of participants with events. | 0 [NA to NA] — NA indicates that upper and lower limit of 90% CI were not estimable due to insufficient number of participants with events. | 50 [NA to NA] — NA indicates that the upper and lower limit of 90% CI were not estimable, as there were insufficient numbers of participants with several participants censored prior to any event.

6. Secondary Outcome: Parts A, B, C, D, F, H, I, J: Clinical Benefit Rate (CBR) as Determined by Investigators/Local Radiologists
Description: CBR was determined by dividing the number of participants who achieved confirmed CR, PR as best overall response (BOR) or stable disease (SD) for ≥24 weeks by the number of participants from the analysis population. CBR was assessed by investigators/local radiologists according to RECIST v1.1. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) had a reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum diameters while on study.
Time Frame: as for outcome 5
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Part A: Amcenestrant 20 mg | Part A: Amcenestrant 150 mg | Part A: Amcenestrant 200 mg | Part A: Amcenestrant 400 mg | Part A: Amcenestrant 600 mg | Part A: Amcenestrant 300 mg BID | Part B: Amcenestrant 400 mg | Part C: Amcenestrant 200 mg + Palbociclib 125 mg | Part C: Amcenestrant 400 mg + Palbociclib 125 mg | Part D: Amcenestrant 200 mg + Palbociclib 125 mg | Part F: Amcenestrant 200 mg + Alpelisib 300 mg | Part H: Amcenestrant 200 mg + Everolimus 5 mg | Part H: Amcenestrant 200 mg + Everolimus 10 mg | Part I: Amcenestrant 200 mg + Everolimus 10 mg | Part J: Amcenestrant 200 mg + Abemaciclib 100 mg BID | Part J: Amcenestrant 200 mg + Abemaciclib 150 mg BID
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 4 | 46 | 9 | 6 | 29 | 7 | 2 | 3 | 1 | 3 | 2
percentage of participants | 0 [NA to NA] — NA indicates that upper and lower limit of 90% CI were not estimable due to insufficient number of participants with events. | 66.7 [13.5 to 98.3] | 75.0 [24.9 to 98.7] | 66.7 [13.5 to 98.3] | 33.3 [1.7 to 86.5] | 25.0 [1.3 to 75.1] | 26.1 [15.8 to 38.8] | 44.4 [16.9 to 74.9] | 50.0 [15.3 to 84.7] | 75.9 [59.4 to 88.1] | 14.3 [NA to NA] — NA indicates that the upper and lower limit of 90% CI were not estimable, as there were insufficient numbers of participants with several participants censored prior to any event. | 50 [NA to NA] — NA indicates that the upper and lower limit of 90% CI were not estimable, as there were insufficient numbers of participants with several participants censored prior to any event. | 33.3 [NA to NA] — NA indicates that the upper and lower limit of 90% CI were not estimable, as there were insufficient numbers of participants with several participants censored prior to any event. | 0 [NA to NA] — NA indicates that upper and lower limit of 90% CI were not estimable due to insufficient number of participants with events. | 66.7 [NA to NA] — NA indicates that the upper and lower limit of 90% CI were not estimable, as there were insufficient numbers of participants with several participants censored prior to any event. | 50 [NA to NA] — NA indicates that the upper and lower limit of 90% CI were not estimable, as there were insufficient numbers of participants with several participants censored prior to any event.

7. Secondary Outcome: Part B: Clinical Benefit Rate as Determined by Independent Central Review
Description: CBR was determined by dividing the number of participants who achieved confirmed CR, PR as BOR or SD for ≥24 weeks by the number of participants from the analysis population. CBR was assessed by ICR according to RECIST v1.1. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) had a reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Part B: Amcenestrant 400 mg
Number analyzed (Participants) | 46
percentage of participants | 28.3 [17.6 to 41.1]

8. Secondary Outcome: Parts A, B, C, D, F, H, I, J: Duration of Response (DOR) as Determined by Investigators/Local Radiologists
Description: DOR was defined as the time interval from the date of the first occurrence of confirmed CR or PR to the date of the first documentation of disease progression or death due to disease progression, whichever occurred first. DOR was assessed by investigators/local radiologists according to RECIST v1.1. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) had a reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study, an absolute increase of at least 5 mm in the sum. Appearance of 1 or more new lesions was also considered progression.
Time Frame: as for outcome 5
Population: The efficacy population included all treated participants with measurable disease at study entry who provided a baseline and at least 1 post-baseline evaluable tumor assessment. Participants with an early progression as per RECIST v1.1 or who died from disease progression were also included in this set. Only participants with CR or PR (responders) were included in the analysis.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Part A: Amcenestrant 20 mg | Part A: Amcenestrant 150 mg | Part A: Amcenestrant 200 mg | Part A: Amcenestrant 400 mg | Part A: Amcenestrant 600 mg | Part A: Amcenestrant 300 mg BID | Part B: Amcenestrant 400 mg | Part C: Amcenestrant 200 mg + Palbociclib 125 mg | Part C: Amcenestrant 400 mg + Palbociclib 125 mg | Part D: Amcenestrant 200 mg + Palbociclib 125 mg | Part F: Amcenestrant 200 mg + Alpelisib 300 mg | Part H: Amcenestrant 200 mg + Everolimus 5 mg | Part H: Amcenestrant 200 mg + Everolimus 10 mg | Part I: Amcenestrant 200 mg + Everolimus 10 mg | Part J: Amcenestrant 200 mg + Abemaciclib 100 mg BID | Part J: Amcenestrant 200 mg + Abemaciclib 150 mg BID
Number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 4 | 2 | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 1
weeks |  | 23.9 [NA to NA] — NA indicates that upper and lower limit of 95% CI could not be calculated for only 1 participant. |  |  |  |  | NA [32.14 to NA] — NA indicates that median and upper limit of 95% CI were not estimable due to insufficient number of participants with events. | 32.2 [24.14 to NA] — NA indicates that upper limit of 95% CI was not estimable due to insufficient number of participants with events. |  | 52.4 [16.00 to NA] — NA indicates that upper limit of 95% CI was not estimable due to insufficient number of participants with events. |  |  |  |  |  | 11.43 [NA to NA] — NA indicates that upper and lower limit of 95% CI could not be calculated for only 1 participant.

9. Secondary Outcome: Part B: Duration of Response as Determined by Independent Central Review
Description: DOR was defined as the time interval from the date of the first occurrence of confirmed CR or PR to the date of the first documentation of disease progression or death due to disease progression, whichever occurred first. DOR was assessed by ICR according to RECIST v1.1. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) had a reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study, an absolute increase of at least 5 mm in the sum. Appearance of 1 or more new lesions was also considered progression.
Time Frame: as for outcome 2
Population: as for outcome 8
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Part B: Amcenestrant 400 mg
Number analyzed (Participants) | 5
weeks | NA [18.71 to NA] — NA indicates that median and upper limit of 95% CI were not estimable due to insufficient number of participants with events.

10. Secondary Outcome: Parts A, B, C, D, F, H, I, J: Progression-Free Survival (PFS) as Determined by Investigators/Local Radiologists
Description: PFS was defined as time from the date of the first treatment intake to the date of the first documentation of objective PD according to RECIST v1.1, clinical PD or death due to any cause, whichever occurred first. PFS was assessed by investigators/local radiologists. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study, an absolute increase of at least 5 mm in the sum. Appearance of 1 or more new lesions was also considered progression.
Time Frame: as for outcome 5
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Part A: Amcenestrant 20 mg | Part A: Amcenestrant 150 mg | Part A: Amcenestrant 200 mg | Part A: Amcenestrant 400 mg | Part A: Amcenestrant 600 mg | Part A: Amcenestrant 300 mg BID | Part B: Amcenestrant 400 mg | Part C: Amcenestrant 200 mg + Palbociclib 125 mg | Part C: Amcenestrant 400 mg + Palbociclib 125 mg | Part D: Amcenestrant 200 mg + Palbociclib 125 mg | Part F: Amcenestrant 200 mg + Alpelisib 300 mg | Part H: Amcenestrant 200 mg + Everolimus 5 mg | Part H: Amcenestrant 200 mg + Everolimus 10 mg | Part I: Amcenestrant 200 mg + Everolimus 10 mg | Part J: Amcenestrant 200 mg + Abemaciclib 100 mg BID | Part J: Amcenestrant 200 mg + Abemaciclib 150 mg BID
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 4 | 46 | 9 | 6 | 29 | 7 | 2 | 3 | 1 | 3 | 2
weeks | 7.3 [6.29 to 15.29] | 31.3 [5.29 to 41.71] | 31.3 [6.14 to 31.57] | 32.3 [8.43 to 90.57] | 7.9 [7.57 to 39.00] | 7.7 [7.14 to 32.00] | 8.3 [7.86 to 23.14] | 44.3 [7.43 to 80.43] | 60.0 [7.43 to NA] — NA indicates that upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 79.7 [40.00 to NA] — NA indicates that upper limit of 95% CI was not estimable due to insufficient number of participants with events. | NA [NA to NA] — NA indicates that median, upper and lower limit of 95% CI were not estimable due to insufficient number of participants with events. | NA [NA to NA] — NA indicates that median, upper and lower limit of 95% CI were not estimable due to insufficient number of participants with events. | NA [NA to NA] — NA indicates that median, upper and lower limit of 95% CI were not estimable due to insufficient number of participants with events. | NA [NA to NA] — NA indicates that median, upper and lower limit of 95% CI were not estimable due to insufficient number of participants with events. | NA [NA to NA] — NA indicates that median, upper and lower limit of 95% CI were not estimable due to insufficient number of participants with events. | NA [NA to NA] — NA indicates that median, upper and lower limit of 95% CI were not estimable due to insufficient number of participants with events.

11. Secondary Outcome: Parts A, B, C, D: Objective Response Rate as Determined by Investigators/Local Radiologists According to Estrogen Receptor 1 (ESR1) Mutation at Baseline
Description: ORR was determined by dividing the number of participants who achieved confirmed CR or PR by the number of participants from the analysis population. ORR was assessed by investigators/local radiologists according to RECIST v1.1. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) had a reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. The ESR1 gene mutation status (mutated or wild-type) was analyzed by multiplex droplet digital polymerase chain reaction (ddPCR) after extraction of plasma circulating deoxyribonucleic acid (DNA). The baseline value was defined as the last value or measurement taken up to the date and time of the first dose of study treatment irrespective of the treatment.
Time Frame: From Baseline (Day 1) up to maximum exposure of study treatment; approximately 90, 278, 140, 228 weeks for Parts A, B, C, D respectively
Population: Analysis was performed on the efficacy population. As pre-specified in statistical analysis plan (SAP), analysis was performed on pooled population [Part A and B: Amcenestrant (Dose >20 mg); Parts C and D: Amcenestrant 200 mg + Palbociclib 125 mg] based on the pharmacodynamic effect to maximize sample size within each arm to provide more robust estimates. Only participants with data collected for each specified category are reported.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Part A and B: Amcenestrant (Dose >20 mg): Participants who received amcenestrant at a dose >20 mg in Parts A and B were included in this cohort.
- Parts C and D: Amcenestrant 200 mg + Palbociclib 125 mg: Participants who received amcenestrant 200 mg along with palbociclib 125 mg in Parts C and D were included in this cohort.
Arm/Group | Part A and B: Amcenestrant (Dose >20 mg) | Parts C and D: Amcenestrant 200 mg + Palbociclib 125 mg
Number analyzed (Participants) | 59 | 38
percentage of participants
  Wild-Type: number analyzed (Participants) | 30 | 27
  Wild-Type | 13.3 [4.7 to 28.0] | 33.3 [18.6 to 50.9]
  Mutated: number analyzed (Participants) | 28 | 11
  Mutated | 3.6 [0.2 to 15.9] | 27.3 [7.9 to 56.4]
  Unknown: number analyzed (Participants) | 1 | 0
  Unknown | 0 [NA to NA] — NA indicates that upper and lower limit of 90% CI were not estimable due to insufficient number of participants with events. |

12. Secondary Outcome: Part B: Objective Response Rate as Determined by Independent Central Review According to Estrogen Receptor 1 Mutation at Baseline
Description: ORR was determined by dividing the number of participants who achieved confirmed CR or PR by the number of participants from the analysis population. ORR was assessed by ICR according to RECIST v1.1. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) had a reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. The ESR1 gene mutation status (mutated or wild-type) was analyzed by multiplex ddPCR after extraction of plasma circulating DNA. The baseline value was defined as the last value or measurement taken up to the date and time of the first dose of study treatment irrespective of the treatment.
Time Frame: Baseline (Day 1) up to maximum exposure of study treatment; approximately 278 weeks
Population: The efficacy population included all treated participants with measurable disease at study entry who provided a baseline and at least 1 post-baseline evaluable tumor assessment. Participants with an early progression as per RECIST v1.1 or who died from disease progression were also included in this set. Only participants with data collected for each specified category are reported.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Part B: Amcenestrant 400 mg
Number analyzed (Participants) | 46
percentage of participants
  Wild-Type: number analyzed (Participants) | 26
  Wild-Type | 15.4 [5.4 to 31.8]
  Mutated: number analyzed (Participants) | 19
  Mutated | 5.3 [0.3 to 22.6]
  Unknown: number analyzed (Participants) | 1
  Unknown | 0 [NA to NA] — NA indicates that upper and lower limit of 90% CI were not estimable due to insufficient number of participants with events.

13. Secondary Outcome: Parts A, B, C, D: Clinical Benefit Rate as Determined by Investigators/Local Radiologists According to Estrogen Receptor 1 Mutation at Baseline
Description: CBR was determined by dividing the number of participants who achieved confirmed CR, PR as BOR or SD for ≥24 weeks by the number of participants from analysis population. CBR was assessed by investigators/local radiologists according to RECIST v1.1. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) had a reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. The ESR1 gene mutation status (mutated or wild-type) was analyzed by multiplex ddPCR after extraction of plasma circulating DNA. Baseline value was defined as the last value or measurement taken up to the date and time of the first dose of study treatment irrespective of the treatment.
Time Frame: as for outcome 11
Population: Analysis was performed on the efficacy population. As pre-specified in SAP, analysis was performed on pooled population [Part A and B: Amcenestrant (Dose >20 mg); Parts C and D: Amcenestrant 200 mg + Palbociclib 125 mg] based on the pharmacodynamic effect to maximize sample size within each arm to provide more robust estimates. Only participants with data collected for each specified category are reported.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Part A and B: Amcenestrant (Dose >20 mg) | Parts C and D: Amcenestrant 200 mg + Palbociclib 125 mg
Number analyzed (Participants) | 59 | 38
percentage of participants
  Wild-Type: number analyzed (Participants) | 30 | 27
  Wild-Type | 36.7 [22.1 to 53.3] | 70.4 [52.9 to 84.3]
  Mutated: number analyzed (Participants) | 28 | 11
  Mutated | 32.1 [17.9 to 49.4] | 63.6 [35.0 to 86.5]
  Unknown: number analyzed (Participants) | 1 | 0
  Unknown | 0 [NA to NA] — NA indicates that upper and lower limit of 90% CI were not estimable due to insufficient number of participants with events. |

14. Secondary Outcome: Parts B, D, I: Time to First Confirmed Response as Determined by Investigators/Local Radiologists
Description: The time to first confirmed response was defined as the time interval from the date of first administration of the study treatment to the date of the first occurrence of confirmed CR or PR. The time to first confirmed response was assessed by investigators/local radiologists according to RECIST v1.1. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) had a reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: as for outcome 5
Population: as for outcome 8
Measure: Median (Full Range); unit: weeks
Arm/Group | Part B: Amcenestrant 400 mg | Part D: Amcenestrant 200 mg + Palbociclib 125 mg | Part I: Amcenestrant 200 mg + Everolimus 10 mg
Number analyzed (Participants) | 4 | 10 | 0
weeks | 8.1 [8 to 40] | 16.2 [8 to 32] |

15. Secondary Outcome: Part B: Time to First Confirmed Response as Determined by Independent Central Review
Description: The time to first confirmed response was defined as the time interval from the date of first administration of the study treatment to the date of the first occurrence of confirmed CR or PR. The time to first confirmed response was assessed by ICR according to RECIST v1.1. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) had a reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: as for outcome 2
Population: as for outcome 8
Measure: Median (Full Range); unit: weeks
Arm/Group | Part B: Amcenestrant 400 mg
Number analyzed (Participants) | 5
weeks | 31.1 [23 to 68]

16. Secondary Outcome: Part A: Number of Participants With 18F-Fluorestradiol Positron Emission Tomography Percentage Reduction
Description: Inhibition of estrogen receptor (ER) occupancy investigation using 18F-FES-PET imaging was a limited invasive procedure that allowed assessment of ER presence by assessing the binding of radiolabeled estradiol, the ligand of ER (signal extinction). Number of participants with percentage reduction (≥90%, ≥70%, ≥50% and ≥30%) in 18F-FES-PET signal are reported. The baseline value was defined as the last value or measurement taken up to the date and time of the first dose of study treatment irrespective of the treatment.
Time Frame: Baseline (within 3 days or more prior to Day 1) and between Day 11 and Day 15 of Cycle 1 (cycle duration=28 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Amcenestrant 20 mg | Part A: Amcenestrant 150 mg | Part A: Amcenestrant 200 mg | Part A: Amcenestrant 400 mg | Part A: Amcenestrant 600 mg | Part A: Amcenestrant 300 mg BID
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 6
Participants
  ≥90% Reduction | 0 | 3 | 2 | 2 | 3 | 2
  ≥70% Reduction | 1 | 3 | 3 | 3 | 3 | 2
  ≥50% Reduction | 1 | 3 | 4 | 3 | 3 | 2
  ≥30% Reduction | 1 | 3 | 4 | 3 | 3 | 3

17. Secondary Outcome: Parts A, B, C, D, H, I, J: Time Interval Between Administration and the Sampling Preceding the First Concentration Above the Lower Limit of Quantification (LLOQ) (Tlag) of Amcenestrant After a Single Oral Administration
Description: Blood samples were collected at the specified timepoint for the measurement of amcenestrant concentrations. Pharmacokinetic (PK) parameters were determined by non-compartmental analysis. LLOQ value for amcenestrant was 5 nanograms per milliliter (ng/mL).
Time Frame: Cycle 1 Day 1 (cycle duration=28 days)
Population: The PK population included all participants from the safety population with at least 1 evaluable treatment concentration after study treatment administration. Only participants with data collected at specified timepoint are reported.
Measure: Median (Full Range); unit: hour
Arm/Group | Part A: Amcenestrant 20 mg | Part A: Amcenestrant 150 mg | Part A: Amcenestrant 200 mg | Part A: Amcenestrant 400 mg | Part A: Amcenestrant 600 mg | Part A: Amcenestrant 300 mg BID | Part B: Amcenestrant 400 mg | Part C: Amcenestrant 200 mg + Palbociclib 125 mg | Part C: Amcenestrant 400 mg + Palbociclib 125 mg | Part D: Amcenestrant 200 mg + Palbociclib 125 mg | Part H: Amcenestrant 200 mg + Everolimus 5 mg | Part H: Amcenestrant 200 mg + Everolimus 10 mg | Part I: Amcenestrant 200 mg + Everolimus 10 mg | Part J: Amcenestrant 200 mg + Abemaciclib 100 mg BID | Part J: Amcenestrant 200 mg + Abemaciclib 150 mg BID
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 6 | 16 | 8 | 6 | 19 | 3 | 3 | 1 | 3 | 2
hour | 0.00 [0.00 to 0.50] | 0.00 [0.00 to 1.58] | 0.00 [0.00 to 0.50] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 1.02] | 0.00 [0.00 to 1.00] | 0.00 [0.00 to 1.00] | 0.470 [0.00 to 1.08] | 0.00 [0.00 to 0.980] | 0.00 [0.00 to 0.980] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]

18. Secondary Outcome: Parts A, B, C, D, H, I, J: Time to Reach Maximum Plasma Concentration (Tmax) of Amcenestrant After a Single Oral Administration
Description: Blood samples were collected at the specified timepoint for the measurement of amcenestrant concentrations. PK parameters were determined by non-compartmental analysis.
Time Frame: Cycle 1 Day 1 (cycle duration=28 days)
Population: as for outcome 17
Measure: Median (Full Range); unit: hour
Arm/Group | Part A: Amcenestrant 20 mg | Part A: Amcenestrant 150 mg | Part A: Amcenestrant 200 mg | Part A: Amcenestrant 400 mg | Part A: Amcenestrant 600 mg | Part A: Amcenestrant 300 mg BID | Part B: Amcenestrant 400 mg | Part C: Amcenestrant 200 mg + Palbociclib 125 mg | Part C: Amcenestrant 400 mg + Palbociclib 125 mg | Part D: Amcenestrant 200 mg + Palbociclib 125 mg | Part H: Amcenestrant 200 mg + Everolimus 5 mg | Part H: Amcenestrant 200 mg + Everolimus 10 mg | Part I: Amcenestrant 200 mg + Everolimus 10 mg | Part J: Amcenestrant 200 mg + Abemaciclib 100 mg BID | Part J: Amcenestrant 200 mg + Abemaciclib 150 mg BID
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 6 | 16 | 8 | 6 | 19 | 3 | 3 | 1 | 3 | 2
hour | 1.52 [1.50 to 2.00] | 3.00 [3.00 to 24.77] | 2.98 [1.98 to 4.02] | 3.00 [1.50 to 3.83] | 3.03 [2.02 to 4.00] | 2.98 [2.00 to 5.95] | 3.98 [1.97 to 9.98] | 5.82 [2.00 to 9.12] | 4.97 [1.00 to 6.13] | 3.03 [2.00 to 23.90] | 4.02 [3.00 to 4.05] | 3.98 [2.00 to 7.92] | 4.00 [4.00 to 4.00] | 3.88 [3.00 to 4.00] | 3.50 [3.00 to 4.00]

19. Secondary Outcome: Parts A, B, C, D, H, I, J: Maximum Plasma Concentration (Cmax) of Amcenestrant After a Single Oral Administration
Description: as for outcome 18
Time Frame: Cycle 1 Day 1 (cycle duration=28 days)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part A: Amcenestrant 20 mg | Part A: Amcenestrant 150 mg | Part A: Amcenestrant 200 mg | Part A: Amcenestrant 400 mg | Part A: Amcenestrant 600 mg | Part A: Amcenestrant 300 mg BID | Part B: Amcenestrant 400 mg | Part C: Amcenestrant 200 mg + Palbociclib 125 mg | Part C: Amcenestrant 400 mg + Palbociclib 125 mg | Part D: Amcenestrant 200 mg + Palbociclib 125 mg | Part H: Amcenestrant 200 mg + Everolimus 5 mg | Part H: Amcenestrant 200 mg + Everolimus 10 mg | Part I: Amcenestrant 200 mg + Everolimus 10 mg | Part J: Amcenestrant 200 mg + Abemaciclib 100 mg BID | Part J: Amcenestrant 200 mg + Abemaciclib 150 mg BID
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 6 | 16 | 8 | 6 | 19 | 3 | 3 | 1 | 3 | 2
ng/mL | 187 (46.7) | 1310 (1380) | 1650 (1340) | 4740 (2920) | 7010 (4180) | 4620 (2740) | 6020 (2810) | 2270 (1130) | 5470 (1280) | 2500 (1110) | 1700 (355) | 1940 (664) | 2330 (NA) — NA indicates that standard deviation (SD) was not estimable for only 1 participant. | 4500 (2860) | 5360 (750)

20. Secondary Outcome: Parts A, B, C, D, H, I, J: Area Under the Plasma Concentration Versus Time Curve From Time Zero to Dosing Interval (AUC0-tau) of Amcenestrant After a Single Oral Administration
Description: Blood samples were collected at the specified timepoint for the measurement of amcenestrant concentrations. PK parameters were determined by non-compartmental analysis. tau=12 h for Part A BID dosing and 24 h for other parts.
Time Frame: Cycle 1 Day 1 (cycle duration=28 days)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Part A: Amcenestrant 20 mg | Part A: Amcenestrant 150 mg | Part A: Amcenestrant 200 mg | Part A: Amcenestrant 400 mg | Part A: Amcenestrant 600 mg | Part A: Amcenestrant 300 mg BID | Part B: Amcenestrant 400 mg | Part C: Amcenestrant 200 mg + Palbociclib 125 mg | Part C: Amcenestrant 400 mg + Palbociclib 125 mg | Part D: Amcenestrant 200 mg + Palbociclib 125 mg | Part H: Amcenestrant 200 mg + Everolimus 5 mg | Part H: Amcenestrant 200 mg + Everolimus 10 mg | Part I: Amcenestrant 200 mg + Everolimus 10 mg | Part J: Amcenestrant 200 mg + Abemaciclib 100 mg BID | Part J: Amcenestrant 200 mg + Abemaciclib 150 mg BID
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 6 | 16 | 8 | 6 | 17 | 3 | 3 | 1 | 3 | 2
ng*h/mL | 1040 (560) | 9140 (8730) | 13600 (13800) | 40400 (17500) | 61100 (36300) | 28200 (16900) | 50900 (26000) | 21300 (5910) | 46400 (4400) | 21400 (10000) | 14100 (3190) | 20900 (4330) | 17900 (NA) — NA indicates that SD was not estimable for only 1 participant. | 36500 (25100) | 38000 (13800)

21. Secondary Outcome: Parts A, B, C, D, F, H, I, J: Time to Reach Maximum Plasma Concentration of Amcenestrant After Repeated Oral Administrations
Description: Blood samples were collected at the specified timepoints for the measurement of amcenestrant concentrations. PK parameters were determined by non-compartmental analysis.
Time Frame: Parts A, B, F, H, I, J: Cycle 1 Day 22; Parts C and D: Cycle 1 Day 21 (cycle duration=28 days)
Population: The PK population included all participants from the safety population with at least 1 evaluable treatment concentration after study treatment administration. Only participants with data collected at specified timepoints are reported.
Measure: Median (Full Range); unit: hour
Arm/Group | Part A: Amcenestrant 20 mg | Part A: Amcenestrant 150 mg | Part A: Amcenestrant 200 mg | Part A: Amcenestrant 400 mg | Part A: Amcenestrant 600 mg | Part A: Amcenestrant 300 mg BID | Part B: Amcenestrant 400 mg | Part C: Amcenestrant 200 mg + Palbociclib 125 mg | Part C: Amcenestrant 400 mg + Palbociclib 125 mg | Part D: Amcenestrant 200 mg + Palbociclib 125 mg | Part F: Amcenestrant 200 mg + Alpelisib 300 mg | Part H: Amcenestrant 200 mg + Everolimus 5 mg | Part H: Amcenestrant 200 mg + Everolimus 10 mg | Part I: Amcenestrant 200 mg + Everolimus 10 mg | Part J: Amcenestrant 200 mg + Abemaciclib 100 mg BID | Part J: Amcenestrant 200 mg + Abemaciclib 150 mg BID
Number analyzed (Participants) | 3 | 2 | 3 | 3 | 3 | 3 | 13 | 8 | 5 | 13 | 3 | 3 | 3 | 1 | 3 | 1
hour | 2.17 [2.00 to 4.02] | 2.97 [2.93 to 3.00] | 2.07 [2.00 to 3.03] | 2.95 [2.02 to 3.78] | 3.00 [3.00 to 4.00] | 2.98 [2.00 to 3.00] | 3.00 [1.02 to 6.00] | 4.88 [1.37 to 8.17] | 4.00 [1.83 to 10.00] | 4.00 [1.75 to 6.00] | 3.22 [1.97 to 3.98] | 2.47 [2.03 to 4.03] | 4.17 [3.95 to 5.92] | 4.07 [4.07 to 4.07] | 2.67 [2.05 to 3.00] | 3.33 [3.33 to 3.33]

22. Secondary Outcome: Parts A, B, C, D, F, H, I, J: Maximum Plasma Concentration of Amcenestrant After Repeated Oral Administrations
Description: as for outcome 21
Time Frame: Parts A, B, F, H, I, J: Cycle 1 Day 22; Parts C and D: Cycle 1 Day 21 (cycle duration=28 days)
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part A: Amcenestrant 20 mg | Part A: Amcenestrant 150 mg | Part A: Amcenestrant 200 mg | Part A: Amcenestrant 400 mg | Part A: Amcenestrant 600 mg | Part A: Amcenestrant 300 mg BID | Part B: Amcenestrant 400 mg | Part C: Amcenestrant 200 mg + Palbociclib 125 mg | Part C: Amcenestrant 400 mg + Palbociclib 125 mg | Part D: Amcenestrant 200 mg + Palbociclib 125 mg | Part F: Amcenestrant 200 mg + Alpelisib 300 mg | Part H: Amcenestrant 200 mg + Everolimus 5 mg | Part H: Amcenestrant 200 mg + Everolimus 10 mg | Part I: Amcenestrant 200 mg + Everolimus 10 mg | Part J: Amcenestrant 200 mg + Abemaciclib 100 mg BID | Part J: Amcenestrant 200 mg + Abemaciclib 150 mg BID
Number analyzed (Participants) | 3 | 2 | 3 | 3 | 3 | 3 | 13 | 8 | 5 | 13 | 3 | 3 | 3 | 1 | 3 | 1
ng/mL | 218 (95.3) | 2390 (1200) | 2150 (873) | 4020 (2460) | 5570 (962) | 5200 (296) | 4380 (1230) | 2060 (831) | 4350 (3190) | 2120 (691) | 4230 (1250) | 3300 (1390) | 2760 (411) | 848 (NA) — NA indicates that SD was not estimable for only 1 participant. | 3350 (1230) | 3820 (NA) — NA indicates that SD was not estimable for only 1 participant.

23. Secondary Outcome: Parts A, B, C, D, F, H, I, J: Area Under the Plasma Concentration Versus Time Curve From Time Zero to Dosing Interval of Amcenestrant After Repeated Oral Administrations
Description: Blood samples were collected at the specified timepoints for the measurement of amcenestrant concentrations. PK parameters were determined by non-compartmental analysis. tau=12 h for Part A BID dosing and 24 h for other parts.
Time Frame: Parts A, B, F, H, I, J: Cycle 1 Day 22; Parts C and D: Cycle 1 Day 21 (cycle duration=28 days)
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Part A: Amcenestrant 20 mg | Part A: Amcenestrant 150 mg | Part A: Amcenestrant 200 mg | Part A: Amcenestrant 400 mg | Part A: Amcenestrant 600 mg | Part A: Amcenestrant 300 mg BID | Part B: Amcenestrant 400 mg | Part C: Amcenestrant 200 mg + Palbociclib 125 mg | Part C: Amcenestrant 400 mg + Palbociclib 125 mg | Part D: Amcenestrant 200 mg + Palbociclib 125 mg | Part F: Amcenestrant 200 mg + Alpelisib 300 mg | Part H: Amcenestrant 200 mg + Everolimus 5 mg | Part H: Amcenestrant 200 mg + Everolimus 10 mg | Part I: Amcenestrant 200 mg + Everolimus 10 mg | Part J: Amcenestrant 200 mg + Abemaciclib 100 mg BID | Part J: Amcenestrant 200 mg + Abemaciclib 150 mg BID
Number analyzed (Participants) | 3 | 2 | 3 | 3 | 3 | 3 | 13 | 8 | 5 | 13 | 3 | 3 | 3 | 1 | 3 | 1
ng*h/mL | 1630 (1120) | 15900 (7350) | 13900 (4380) | 36800 (23500) | 42700 (11200) | 36500 (7680) | 43200 (16200) | 20600 (7520) | 33100 (11400) | 17600 (7540) | 30600 (11900) | 28300 (21100) | 25000 (7180) | 8270 (NA) — NA indicates that SD was not estimable for only 1 participant. | 26600 (12900) | 30300 (NA) — NA indicates that SD was not estimable for only 1 participant.

24. Secondary Outcome: Parts A, B, C, D, F, H, I, J: Plasma Concentration Observed Before Treatment Administration (Ctrough) of Amcenestrant
Description: Blood samples were collected at the specified timepoints for the measurement of amcenestrant concentrations.
Time Frame: Cycle 1: Pre-dose (0 hour) on Day 8 (Parts A, B, C, D), Day 15 (Parts B, C, D), Day 21 (Parts C and D) and Day 22 (Parts A, B, F, H, I, J) (cycle duration=28 days)
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part A: Amcenestrant 20 mg | Part A: Amcenestrant 150 mg | Part A: Amcenestrant 200 mg | Part A: Amcenestrant 400 mg | Part A: Amcenestrant 600 mg | Part A: Amcenestrant 300 mg BID | Part B: Amcenestrant 400 mg | Part C: Amcenestrant 200 mg + Palbociclib 125 mg | Part C: Amcenestrant 400 mg + Palbociclib 125 mg | Part D: Amcenestrant 200 mg + Palbociclib 125 mg | Part F: Amcenestrant 200 mg + Alpelisib 300 mg | Part H: Amcenestrant 200 mg + Everolimus 5 mg | Part H: Amcenestrant 200 mg + Everolimus 10 mg | Part I: Amcenestrant 200 mg + Everolimus 10 mg | Part J: Amcenestrant 200 mg + Abemaciclib 100 mg BID | Part J: Amcenestrant 200 mg + Abemaciclib 150 mg BID
Number analyzed (Participants) | 2 | 1 | 4 | 3 | 3 | 4 | 39 | 7 | 5 | 28 | 3 | 3 | 3 | 1 | 3 | 1
ng/mL
  Cycle 1 Day 8: number analyzed (Participants) | 1 | 1 | 4 | 1 | 1 | 4 | 39 | 7 | 4 | 21 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 1 Day 8 | 0 (NA) — NA indicates that SD was not estimable for only 1 participant. | 91.4 (NA) — NA indicates that SD was not estimable for only 1 participant. | 159 (35.8) | 871 (NA) — NA indicates that SD was not estimable for only 1 participant. | 302 (NA) — NA indicates that SD was not estimable for only 1 participant. | 2220 (1100) | 665 (581) | 348 (180) | 389 (234) | 303 (294) |  |  |  |  |  |
  Cycle 1 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 34 | 6 | 4 | 20 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 1 Day 15 |  |  |  |  |  |  | 553 (605) | 328 (168) | 243 (151) | 226 (198) |  |  |  |  |  |
  Cycle 1 Day 21: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 5 | 28 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 1 Day 21 |  |  |  |  |  |  |  | 359 (132) | 297 (144) | 223 (187) |  |  |  |  |  |
  Cycle 1 Day 22: number analyzed (Participants) | 2 | 1 | 3 | 3 | 3 | 2 | 38 | 0 | 0 | 0 | 3 | 3 | 3 | 1 | 3 | 1
  Cycle 1 Day 22 | 6.80 (9.62) | 75.1 (NA) — NA indicates that SD was not estimable for only 1 participant. | 76.1 (56.0) | 388 (327) | 348 (197) | 1510 (1030) | 598 (460) |  |  |  | 410 (449) | 326 (216) | 346 (128) | 114 (NA) — NA indicates that SD was not estimable for only 1 participant. | 214 (138) | 229 (NA) — NA indicates that SD was not estimable for only 1 participant.

25. Secondary Outcome: Part B: Cumulated Amount of Amcenestrant Excreted in Urine From Time 0 to 24 Hours (Ae0-24)
Description: Urine samples were collected at the specified timepoints for the measurement of amcenestrant amount excreted in urine.
Time Frame: Day 22 of Cycle 1 (cycle duration=28 days)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ng
Arm/Group | Part B: Amcenestrant 400 mg
Number analyzed (Participants) | 9
ng | 30800 (36100)

26. Secondary Outcome: Part A (QD Regimen): Geometric Mean Ratio of Area Under the Plasma Concentration Versus Time Curve From Time Zero to 24 Hours (AUC0-24) of Amcenestrant
Description: The food effect was assessed by comparing the geometric means of AUC0-24 between Cycle 1 Day 1 (fasted condition) and Cycle 1 Day 3 (fed condition) in Part A.
Time Frame: Days 1 and 3 of Cycle 1 (cycle duration=28 days)
Population: The food-effect population included participants who received study treatment in fed condition on Cycle 1 Day 3 and in fasted condition on Cycle 1 Day 1 in Part A. As pre-specified in SAP, food effect was assessed in Part A QD regimen cohorts only.
Measure: Number (90% Confidence Interval); unit: ratio
Arm/Group | Part A: Amcenestrant 20 mg | Part A: Amcenestrant 150 mg | Part A: Amcenestrant 200 mg | Part A: Amcenestrant 400 mg | Part A: Amcenestrant 600 mg
Number analyzed (Participants) | 2 | 1 | 4 | 1 | 3
ratio | 1.05 [0.60 to 1.83] | 0.69 [0.31 to 1.50] | 1.77 [1.20 to 2.62] | 1.12 [0.51 to 2.45] | 1.38 [0.88 to 2.17]

27. Secondary Outcome: Part A (QD Regimen): Geometric Mean Ratio of Maximum Plasma Concentration of Amcenestrant
Description: The food effect was assessed by comparing the geometric means of Cmax between Cycle 1 Day 1 (fasted condition) and Cycle 1 Day 3 (fed condition) in Part A.
Time Frame: Days 1 and 3 of Cycle 1 (cycle duration=28 days)
Population: as for outcome 26
Measure: Number (90% Confidence Interval); unit: ratio
Arm/Group | Part A: Amcenestrant 20 mg | Part A: Amcenestrant 150 mg | Part A: Amcenestrant 200 mg | Part A: Amcenestrant 400 mg | Part A: Amcenestrant 600 mg
Number analyzed (Participants) | 2 | 1 | 4 | 1 | 3
ratio | 0.80 [0.41 to 1.58] | 0.41 [0.16 to 1.07] | 1.67 [1.04 to 2.69] | 1.38 [0.53 to 3.59] | 1.43 [0.83 to 2.48]

28. Secondary Outcome: Parts C and D: Time to Reach Maximum Plasma Concentration of Palbociclib After First Dose and Repeated Oral Administrations in Combination With Amcenestrant
Description: Blood samples were collected after single dose (Day 1) and repeated oral administrations (Day 21) of palbociclib in combination with amcenestrant for the measurement of palbociclib concentrations. PK parameters were determined by non-compartmental analysis.
Time Frame: Days 1 and 21 of Cycle 1 (cycle duration=28 days)
Population: as for outcome 21
Measure: Median (Full Range); unit: hour
Arm/Group | Part C: Amcenestrant 200 mg + Palbociclib 125 mg | Part C: Amcenestrant 400 mg + Palbociclib 125 mg | Part D: Amcenestrant 200 mg + Palbociclib 125 mg
Number analyzed (Participants) | 8 | 6 | 19
hour
  Cycle 1 Day 1 | 5.70 [3.00 to 10.00] | 3.99 [2.02 to 7.98] | 6.00 [2.07 to 24.00]
  Cycle 1 Day 21: number analyzed (Participants) | 8 | 5 | 13
  Cycle 1 Day 21 | 4.10 [1.93 to 9.97] | 6.00 [3.02 to 8.08] | 4.75 [3.00 to 9.58]

29. Secondary Outcome: Parts C and D: Maximum Plasma Concentration of Palbociclib After First Dose and Repeated Oral Administrations in Combination With Amcenestrant
Description: Blood samples were collected after single dose (Day 1) and repeated oral administrations (Day 21) of palbociclib in combination with amcenestrant. PK parameters were determined by non-compartmental analysis.
Time Frame: Days 1 and 21 of Cycle 1 (cycle duration=28 days)
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part C: Amcenestrant 200 mg + Palbociclib 125 mg | Part C: Amcenestrant 400 mg + Palbociclib 125 mg | Part D: Amcenestrant 200 mg + Palbociclib 125 mg
Number analyzed (Participants) | 8 | 6 | 19
ng/mL
  Cycle 1 Day 1 | 70.4 (26.1) | 64.7 (28.4) | 62.3 (17.5)
  Cycle 1 Day 21: number analyzed (Participants) | 8 | 5 | 13
  Cycle 1 Day 21 | 98.1 (37.6) | 59.4 (28.1) | 96.3 (34.9)

30. Secondary Outcome: Parts C and D: Area Under the Plasma Concentration Versus Time Curve From Time Zero to 24 Hours of Palbociclib After First Dose and Repeated Oral Administrations in Combination With Amcenestrant
Description: as for outcome 29
Time Frame: Days 1 and 21 of Cycle 1 (cycle duration=28 days)
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Part C: Amcenestrant 200 mg + Palbociclib 125 mg | Part C: Amcenestrant 400 mg + Palbociclib 125 mg | Part D: Amcenestrant 200 mg + Palbociclib 125 mg
Number analyzed (Participants) | 8 | 6 | 19
ng*h/mL
  Cycle 1 Day 1 | 1040 (257) | 889 (376) | 949 (265)
  Cycle 1 Day 21: number analyzed (Participants) | 8 | 5 | 13
  Cycle 1 Day 21 | 1660 (751) | 823 (266) | 1570 (523)

31. Secondary Outcome: Part F: Time to Reach Maximum Plasma Concentration of Alpelisib After Repeated Oral Administrations Alone or in Combination With Amcenestrant
Description: Blood samples were collected after 3-day repeated oral administrations of alpelisib as monotherapy (Day 3) and after 22-day repeated oral administrations of alpelisib in combination with repeated doses of amcenestrant (Day 22). PK parameters were determined by non-compartmental analysis.
Time Frame: Days 3 and 22 of Cycle 1 (cycle duration=28 days)
Population: as for outcome 21
Measure: Median (Full Range); unit: hour
Arm/Group | Part F: Amcenestrant 200 mg + Alpelisib 300 mg
Number analyzed (Participants) | 7
hour
  Cycle 1 Day 3 | 3.02 [1.02 to 9.00]
  Cycle 1 Day 22: number analyzed (Participants) | 2
  Cycle 1 Day 22 | 1.69 [1.25 to 2.12]

32. Secondary Outcome: Part F: Maximum Plasma Concentration of Alpelisib After Repeated Oral Administrations Alone or in Combination With Amcenestrant
Description: as for outcome 31
Time Frame: Days 3 and 22 of Cycle 1 (cycle duration=28 days)
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part F: Amcenestrant 200 mg + Alpelisib 300 mg
Number analyzed (Participants) | 7
ng/mL
  Cycle 1 Day 3 | 2430 (631)
  Cycle 1 Day 22: number analyzed (Participants) | 2
  Cycle 1 Day 22 | 3480 (516)

33. Secondary Outcome: Part F: Area Under the Plasma Concentration Versus Time Curve From Time Zero to 24 Hours of Alpelisib After Repeated Oral Administrations Alone or in Combination With Amcenestrant
Description: as for outcome 31
Time Frame: Days 3 and 22 of Cycle 1 (cycle duration=28 days)
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Part F: Amcenestrant 200 mg + Alpelisib 300 mg
Number analyzed (Participants) | 7
ng*h/mL
  Cycle 1 Day 3 | 28700 (7890)
  Cycle 1 Day 22: number analyzed (Participants) | 2
  Cycle 1 Day 22 | 27300 (6910)

34. Secondary Outcome: Parts H and I: Time to Reach Maximum Plasma Concentration of Everolimus After First Dose and Repeated Oral Administrations in Combination With Amcenestrant
Description: Blood samples were collected after single dose (Day 1) and repeated oral administrations (Day 22) of everolimus in combination with amcenestrant. PK parameters were determined by non-compartmental analysis.
Time Frame: Days 1 and 22 of Cycle 1 (cycle duration=28 days)
Population: The PK population included all participants from the safety population with at least 1 evaluable treatment concentration after study treatment administration.
Measure: Median (Full Range); unit: hour
Arm/Group | Part H: Amcenestrant 200 mg + Everolimus 5 mg | Part H: Amcenestrant 200 mg + Everolimus 10 mg | Part I: Amcenestrant 200 mg + Everolimus 10 mg
Number analyzed (Participants) | 3 | 3 | 1
hour
  Cycle 1 Day 1 | 1.02 [1.00 to 3.00] | 2.00 [0.98 to 3.02] | 1.00 [1.00 to 1.00]
  Cycle 1 Day 22 | 1.00 [0.97 to 1.47] | 2.08 [0.98 to 3.03] | 1.10 [1.10 to 1.10]

35. Secondary Outcome: Parts H and I: Maximum Plasma Concentration of Everolimus After First Dose and Repeated Oral Administrations in Combination With Amcenestrant
Description: as for outcome 34
Time Frame: Days 1 and 22 of Cycle 1 (cycle duration=28 days)
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part H: Amcenestrant 200 mg + Everolimus 5 mg | Part H: Amcenestrant 200 mg + Everolimus 10 mg | Part I: Amcenestrant 200 mg + Everolimus 10 mg
Number analyzed (Participants) | 3 | 3 | 1
ng/mL
  Cycle 1 Day 1 | 38.7 (21.9) | 64.8 (3.54) | 43.5 (NA) — NA indicates that SD was not estimable for only 1 participant.
  Cycle 1 Day 22 | 24.4 (6.32) | 37.6 (15.5) | 46.7 (NA) — NA indicates that SD was not estimable for only 1 participant.

36. Secondary Outcome: Parts H and I: Area Under the Plasma Concentration Versus Time Curve From Time Zero to 24 Hours of Everolimus After First Dose and Repeated Oral Administrations in Combination With Amcenestrant
Description: as for outcome 34
Time Frame: Days 1 and 22 of Cycle 1 (cycle duration=28 days)
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Part H: Amcenestrant 200 mg + Everolimus 5 mg | Part H: Amcenestrant 200 mg + Everolimus 10 mg | Part I: Amcenestrant 200 mg + Everolimus 10 mg
Number analyzed (Participants) | 3 | 3 | 1
ng*h/mL
  Cycle 1 Day 1 | 210 (117) | 381 (159) | 246 (NA) — NA indicates that SD was not estimable for only 1 participant.
  Cycle 1 Day 22 | 144 (35.0) | 319 (156) | 295 (NA) — NA indicates that SD was not estimable for only 1 participant.

37. Secondary Outcome: Part J: Time to Reach Maximum Plasma Concentration of Abemaciclib and Its Metabolites M2, M18 and M20 After First Dose and Repeated Oral Administrations in Combination With Amcenestrant
Description: Blood samples were collected after single dose (Day 1) and repeated oral administrations (Day 22) of abemaciclib in combination with amcenestrant. PK parameters were determined by non-compartmental analysis.
Time Frame: Days 1 and 22 of Cycle 1 (cycle duration=28 days)
Population: as for outcome 21
Measure: Median (Full Range); unit: hour
Arm/Group | Part J: Amcenestrant 200 mg + Abemaciclib 100 mg BID | Part J: Amcenestrant 200 mg + Abemaciclib 150 mg BID
Number analyzed (Participants) | 3 | 2
hour
  Abemaciclib: Cycle 1 Day 1 | 5.75 [3.00 to 9.00] | 6.00 [4.00 to 8.00]
  Abemaciclib: Cycle 1 Day 22: number analyzed (Participants) | 3 | 1
  Abemaciclib: Cycle 1 Day 22 | 3.00 [2.67 to 4.03] | 8.00 [8.00 to 8.00]
  M2: Cycle 1 Day 1 | 3.88 [3.00 to 4.00] | 6.50 [4.00 to 9.00]
  M2: Cycle 1 Day 22: number analyzed (Participants) | 3 | 1
  M2: Cycle 1 Day 22 | 2.67 [1.03 to 3.00] | 4.00 [4.00 to 4.00]
  M18: Cycle 1 Day 1 | 4.00 [3.88 to 8.00] | 8.00 [8.00 to 8.00]
  M18: Cycle 1 Day 22: number analyzed (Participants) | 3 | 1
  M18: Cycle 1 Day 22 | 2.67 [1.97 to 4.00] | 4.00 [4.00 to 4.00]
  M20: Cycle 1 Day 1 | 8.07 [3.00 to 9.00] | 8.50 [8.00 to 9.00]
  M20: Cycle 1 Day 22: number analyzed (Participants) | 3 | 1
  M20: Cycle 1 Day 22 | 1.03 [0.00 to 4.67] | 8.67 [8.67 to 8.67]

38. Secondary Outcome: Part J: Maximum Plasma Concentration of Abemaciclib and Its Metabolites M2, M18 and M20 After First Dose and Repeated Oral Administrations in Combination With Amcenestrant
Description: as for outcome 37
Time Frame: Days 1 and 22 of Cycle 1 (cycle duration=28 days)
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part J: Amcenestrant 200 mg + Abemaciclib 100 mg BID | Part J: Amcenestrant 200 mg + Abemaciclib 150 mg BID
Number analyzed (Participants) | 3 | 2
ng/mL
  Abemaciclib: Cycle 1 Day 1 | 91.6 (58.4) | 152 (44.5)
  Abemaciclib: Cycle 1 Day 22: number analyzed (Participants) | 3 | 1
  Abemaciclib: Cycle 1 Day 22 | 109 (45.6) | 87.8 (NA) — NA indicates that SD was not estimable for only 1 participant.
  M2: Cycle 1 Day 1 | 17.8 (3.46) | 55.3 (22.0)
  M2: Cycle 1 Day 22: number analyzed (Participants) | 3 | 1
  M2: Cycle 1 Day 22 | 69.1 (20.5) | 106 (NA) — NA indicates that SD was not estimable for only 1 participant.
  M18: Cycle 1 Day 1 | 6.37 (0.514) | 22.0 (4.24)
  M18: Cycle 1 Day 22: number analyzed (Participants) | 3 | 1
  M18: Cycle 1 Day 22 | 35.1 (17.2) | 89.5 (NA) — NA indicates that SD was not estimable for only 1 participant.
  M20: Cycle 1 Day 1 | 31.2 (2.84) | 65.5 (8.13)
  M20: Cycle 1 Day 22: number analyzed (Participants) | 3 | 1
  M20: Cycle 1 Day 22 | 100 (17.3) | 153 (NA) — NA indicates that SD was not estimable for only 1 participant.

39. Secondary Outcome: Part J: Area Under the Plasma Concentration Versus Time Curve From Time Zero to 12 Hours of Abemaciclib and Its Metabolites M2, M18 and M20 After First Dose and Repeated Oral Administrations in Combination With Amcenestrant
Description: as for outcome 37
Time Frame: Days 1 and 22 of Cycle 1 (cycle duration=28 days)
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Part J: Amcenestrant 200 mg + Abemaciclib 100 mg BID | Part J: Amcenestrant 200 mg + Abemaciclib 150 mg BID
Number analyzed (Participants) | 3 | 2
ng*h/mL
  Abemaciclib: Cycle 1 Day 1: number analyzed (Participants) | 2 | 2
  Abemaciclib: Cycle 1 Day 1 | 994 (700) | 1330 (478)
  Abemaciclib: Cycle 1 Day 22: number analyzed (Participants) | 3 | 0
  Abemaciclib: Cycle 1 Day 22 | 1050 (532) |
  M2: Cycle 1 Day 1: number analyzed (Participants) | 2 | 1
  M2: Cycle 1 Day 1 | 160 (45.0) | 554 (NA) — NA indicates that SD was not estimable for only 1 participant.
  M2: Cycle 1 Day 22: number analyzed (Participants) | 3 | 1
  M2: Cycle 1 Day 22 | 610 (170) | 1130 (NA) — NA indicates that SD was not estimable for only 1 participant.
  M18: Cycle 1 Day 1: number analyzed (Participants) | 2 | 1
  M18: Cycle 1 Day 1 | 47.6 (0.468) | 218 (NA) — NA indicates that SD was not estimable for only 1 participant.
  M18: Cycle 1 Day 22: number analyzed (Participants) | 3 | 1
  M18: Cycle 1 Day 22 | 314 (141) | 926 (NA) — NA indicates that SD was not estimable for only 1 participant.
  M20: Cycle 1 Day 1: number analyzed (Participants) | 2 | 0
  M20: Cycle 1 Day 1 | 295 (9.12) |
  M20: Cycle 1 Day 22: number analyzed (Participants) | 3 | 0
  M20: Cycle 1 Day 22 | 997 (219) |

40. Secondary Outcome: Parts A, B, J: Post/Pre--Treatment Ratio of 4 Beta (β)-Hydroxycholesterol
Description: Ratios of 4β-hydroxycholesterol concentrations were calculated from plasma samples collected before and after amcenestrant administration.
Time Frame: Pre-treatment on Day 1 of Cycle 1; post-treatment on Day 22 of Cycle 1, Day 1 and Day 28 (only for Part J) of Cycle 2 (cycle duration=28 days)
Population: The PK population included all participants from the safety population with at least 1 evaluable treatment concentration after study treatment administration. Only participants with data collected at specified timepoints are reported. The study was terminated prior to data collection for Part J for this outcome measure.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Part A: Amcenestrant 20 mg | Part A: Amcenestrant 150 mg | Part A: Amcenestrant 200 mg | Part A: Amcenestrant 400 mg | Part A: Amcenestrant 600 mg | Part A: Amcenestrant 300 mg BID | Part B: Amcenestrant 400 mg | Part J: Amcenestrant 200 mg + Abemaciclib 100 mg BID | Part J: Amcenestrant 200 mg + Abemaciclib 150 mg BID
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 2 | 3 | 13 | 0 | 0
ratio
  Cycle 1 Day 22/Cycle 1 Day 1: number analyzed (Participants) | 2 | 2 | 3 | 3 | 2 | 2 | 13 | 0 | 0
  Cycle 1 Day 22/Cycle 1 Day 1 | 0.817 (0.168) | 1.18 (0.294) | 1.29 (0.263) | 1.61 (0.336) | 2.24 (1.29) | 2.17 (0.377) | 1.68 (0.577) |  |
  Cycle 2 Day 1/Cycle 1 Day 1: number analyzed (Participants) | 3 | 3 | 4 | 3 | 2 | 3 | 12 | 0 | 0
  Cycle 2 Day 1/Cycle 1 Day 1 | 1.09 (0.304) | 1.13 (0.432) | 1.39 (0.207) | 1.83 (0.569) | 2.40 (0.559) | 2.99 (1.58) | 1.89 (0.627) |  |
  Cycle 2 Day 28/Cycle 1 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment administration (Day 1) up to 30 days after the last dose of study treatment administration; approximately 94, 282, 144, 232, 96, 59, 11, 130 weeks for Parts A, B, C, D, F, H, I, J respectively. All-cause mortality (deaths) were collected from first dose of study treatment administration (Day 1) to the end of follow-up for death for each participant; up to approximately 372 weeks
Description: Analysis was performed on the safety population.
Arm/Group | Part A: Amcenestrant 20 mg | Part A: Amcenestrant 150 mg | Part A: Amcenestrant 200 mg | Part A: Amcenestrant 400 mg | Part A: Amcenestrant 600 mg | Part A: Amcenestrant 300 mg BID | Part B: Amcenestrant 400 mg | Part C: Amcenestrant 200 mg + Palbociclib 125 mg | Part C: Amcenestrant 400 mg + Palbociclib 125 mg | Part D: Amcenestrant 200 mg + Palbociclib 125 mg | Part F: Amcenestrant 200 mg + Alpelisib 300 mg | Part H: Amcenestrant 200 mg + Everolimus 5 mg | Part H: Amcenestrant 200 mg + Everolimus 10 mg | Part I: Amcenestrant 200 mg + Everolimus 10 mg | Part J: Amcenestrant 200 mg + Abemaciclib 100 mg BID | Part J: Amcenestrant 200 mg + Abemaciclib 150 mg BID
All-Cause Mortality (participants affected / at risk) | 1/3 | 1/3 | 0/4 | 0/3 | 1/3 | 0/6 | 4/49 | 1/9 | 0/6 | 0/30 | 2/8 | 0/3 | 0/3 | 0/1 | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/3 | 1/4 | 0/3 | 1/3 | 3/6 | 15/49 | 2/9 | 1/6 | 8/30 | 6/8 | 1/3 | 0/3 | 1/1 | 0/3 | 1/2
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 4/4 | 3/3 | 3/3 | 6/6 | 49/49 | 9/9 | 6/6 | 29/30 | 8/8 | 3/3 | 3/3 | 1/1 | 3/3 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Amcenestrant 20 mg (N=3) | Part A: Amcenestrant 150 mg (N=3) | Part A: Amcenestrant 200 mg (N=4) | Part A: Amcenestrant 400 mg (N=3) | Part A: Amcenestrant 600 mg (N=3) | Part A: Amcenestrant 300 mg BID (N=6) | Part B: Amcenestrant 400 mg (N=49) | Part C: Amcenestrant 200 mg + Palbociclib 125 mg (N=9) | Part C: Amcenestrant 400 mg + Palbociclib 125 mg (N=6) | Part D: Amcenestrant 200 mg + Palbociclib 125 mg (N=30) | Part F: Amcenestrant 200 mg + Alpelisib 300 mg (N=8) | Part H: Amcenestrant 200 mg + Everolimus 5 mg (N=3) | Part H: Amcenestrant 200 mg + Everolimus 10 mg (N=3) | Part I: Amcenestrant 200 mg + Everolimus 10 mg (N=1) | Part J: Amcenestrant 200 mg + Abemaciclib 100 mg BID (N=3) | Part J: Amcenestrant 200 mg + Abemaciclib 150 mg BID (N=2)
Breast Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional State (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine With Aura (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient Ischaemic Attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal Detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial Effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Superior Vena Cava Syndrome (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Duodenal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema Mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaundice Cholestatic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disease Progression (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acetabulum Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Amcenestrant 20 mg (N=3) | Part A: Amcenestrant 150 mg (N=3) | Part A: Amcenestrant 200 mg (N=4) | Part A: Amcenestrant 400 mg (N=3) | Part A: Amcenestrant 600 mg (N=3) | Part A: Amcenestrant 300 mg BID (N=6) | Part B: Amcenestrant 400 mg (N=49) | Part C: Amcenestrant 200 mg + Palbociclib 125 mg (N=9) | Part C: Amcenestrant 400 mg + Palbociclib 125 mg (N=6) | Part D: Amcenestrant 200 mg + Palbociclib 125 mg (N=30) | Part F: Amcenestrant 200 mg + Alpelisib 300 mg (N=8) | Part H: Amcenestrant 200 mg + Everolimus 5 mg (N=3) | Part H: Amcenestrant 200 mg + Everolimus 10 mg (N=3) | Part I: Amcenestrant 200 mg + Everolimus 10 mg (N=1) | Part J: Amcenestrant 200 mg + Abemaciclib 100 mg BID (N=3) | Part J: Amcenestrant 200 mg + Abemaciclib 150 mg BID (N=2)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 6 (6) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral Herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 5 (9) | 1 (1) | 1 (1) | 5 (5) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal Mycotic Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases To Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seborrhoeic Keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (8) | 1 (3) | 13 (42) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 1 (2) | 7 (7) | 0 (0) | 2 (2) | 1 (1) | 3 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Polydipsia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed Mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nightmare (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Burning Sensation (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 2 (3) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 6 (8) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (3) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Memory Impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Morton's Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy Peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parkinson's Disease (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry Eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ectropion (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye Irritation (Eye disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye Oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye Pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meibomianitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision Blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meniere's Disease (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot Flush (Vascular disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 7 (7) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jugular Vein Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subclavian Vein Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Varicose Vein (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 1 (1) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 1 (1) | 6 (6) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper-Airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 11 (11) | 2 (2) | 2 (2) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 6 (8) | 3 (4) | 1 (1) | 6 (13) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal Erythema (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal Incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphthous Ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 14 (18) | 2 (3) | 0 (0) | 5 (8) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (5) | 2 (3) | 3 (3) | 0 (0) | 3 (4) | 8 (8) | 1 (1) | 3 (7) | 8 (16) | 6 (9) | 1 (1) | 2 (4) | 1 (1) | 2 (4) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperaesthesia Teeth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intra-Abdominal Haematoma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 11 (13) | 4 (6) | 1 (1) | 8 (13) | 5 (5) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema Mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Teeth Brittle (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (4) | 14 (26) | 3 (4) | 1 (1) | 5 (7) | 3 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic Cytolysis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis Exfoliative Generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 6 (6) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mechanical Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail Disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Night Sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain Of Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 6 (7) | 2 (6) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash Pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin Fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin Irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Xeroderma (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 1 (2) | 1 (1) | 1 (1) | 1 (1) | 10 (12) | 2 (5) | 2 (2) | 8 (15) | 1 (4) | 1 (1) | 3 (6) | 0 (0) | 1 (2) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (3) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteonecrosis Of Jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 2 (2) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain In Jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Temporomandibular Pain And Dysfunction Syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Micturition Urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oliguria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal Pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary Incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Discomfort (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast Mass (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast Pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal Dryness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 9 (9) | 3 (3) | 1 (5) | 4 (7) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Axillary Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Complication Associated With Device (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Face Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 12 (12) | 2 (3) | 1 (1) | 12 (14) | 2 (4) | 2 (4) | 2 (3) | 1 (1) | 2 (2) | 0 (0)
Hyperthermia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza Like Illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal Inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (5) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema Peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Alkaline Phosphatase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Bilirubin Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram Qt Prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-Glutamyltransferase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil Count Abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil Count Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thermal Burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Sponsor decision to prematurely stop the study, it was not linked to any safety concern.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2021-12-08): https://cdn.clinicaltrials.gov/large-docs/57/NCT03284957/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-27): https://cdn.clinicaltrials.gov/large-docs/57/NCT03284957/SAP_001.pdf